CLINICAL TRIAL: NCT00060905
Title: An Inpatient Study of the Effectiveness and Safety of Depakote ER in the Treatment of Mania/Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-540
Record Dates: First submitted 2003-05-15; First posted 2003-05-16 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2006-08

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder (manic or mixed type)
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Valproic Acid

INTERVENTIONS:
Drug: Divalproex Sodium (Depakote ER)

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of Depakote ER compared to placebo in the treatment of bipolar disorder, manic or mixed type in adults.

ELIGIBILITY:
INCLUSION CRITERIA

* Current primary diagnosis of bipolar I disorder, mania or mixed type
* Acute exacerbation of mania associated with bipolar disorder as defined by Mania Rating Scale score >= 18
* Hospitalized no more than 7 days at time of Screening or in process of being admitted
* History of at least one prior manic or mixed episode within past 3 years, exclusive of the current episode. Prior manic or mixed episode must be separated from current episode by at least 2 months of sustained improvement

EXCLUSION CRITERIA

* History of schizophrenia or schizoaffective disorder
* Axis I (e.g., anxiety disorder), or Axis II (e.g., personality disorder) that would interfere with compliance or confound interpretation of study results
* Current manic or mixed episode is drug-induced or secondary to a medical disorder (e.g., AIDS, corticosteroids)
* Current manic or mixed episode is believed to be caused by antidepressant use (i.e., antidepressant-induced mania)
* Had first manic episode after age 60
* Has ever taken clozapine
* Has received depot neuroleptic medication within one inter-injection interval of first dose of study drug
* Urine toxicology screen is positive for phencyclidine (PCP), opiates, cocaine or amphetamines
* History of active alcohol or substance dependence within past 3 months.
* History of failed treatment on adequate valproate therapy for bipolar disorder
* Has taken Depakote (DR or ER) regularly over the last 30 days
* Has serious violent, homicidal, or suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370
Dates: Start 2003-01

PRIMARY OUTCOMES:
Change from baseline to the final evaluation for the MRS from the SADS-C for the intent-to-treat dataset.

SECONDARY OUTCOMES:
Change from baseline to the final evaluation for the Manic Syndrome Scale (MSS), Behavior and Ideation Scale (BIS),
BPRS (and published subscales), Global Assessment Scale (GAS), the Nursing Observation Scale for Inpatient Evaluation (NOSIE), and Burden Questionnaire, as well as the percentage of subjects with at least 50% improvement on the MRS.

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information - Abbott, Study Director — Abbott
Locations (18):
- United States (18):
  - Comprehensive Neuroscience of SCA, Cerritos, California
  - AVI Clinical Research, Torrance, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Mark Lerman, MD, Hoffman Estates, Illinois
  - University of Louisville Bipolar Research Program, Louisville, Kentucky
  - Brentwood Research Inst., Shreveport, Louisiana
  - Centers for Behavioral Health, LLC, Rockville, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Pioneer Research, Baltimore, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Steven A. Glass, MD, Clementon, New Jersey
  - The Holliswood Hospital, Holliswood, New York
  - NYU School of Medicine - Bellevue, New York, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - UT Mental Sciences Institute, Houston, Texas
  - San Antonio State Hospital, San Antonio, Texas
  - CNS of Northern Virginia, Falls Church, Virginia
  - VAMC, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Hirschfeld RM, Bowden CL, Vigna NV, Wozniak P, Collins M. A randomized, placebo-controlled, multicenter study of divalproex sodium extended-release in the acute treatment of mania. J Clin Psychiatry. 2010 Apr;71(4):426-32. doi: 10.4088/JCP.08m04960yel. Epub 2010 Mar 9. PMID 20361904
- [Derived] Bowden CL, Swann AC, Calabrese JR, Rubenfaer LM, Wozniak PJ, Collins MA, Abi-Saab W, Saltarelli M; Depakote ER Mania Study Group. A randomized, placebo-controlled, multicenter study of divalproex sodium extended release in the treatment of acute mania. J Clin Psychiatry. 2006 Oct;67(10):1501-10. doi: 10.4088/jcp.v67n1003. PMID 17107240